CLINICAL TRIAL: NCT04798430
Title: Open-Label Extension Phase 3 Study to Evaluate the Long-Term Efficacy and Safety of LIB003 in Patients With HoFH and HeFH, CVD, or at High Risk for CVD, on Stable Lipid-Lowering Therapy Requiring Additional LDL-C Reduction
Brief Title: Long-term Efficacy and Safety of OLE LIB003 in HoFH, HeFH, and High-risk CVD Patients Requiring Further LDL-C Reduction
Acronym: LIBerate-OLE
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: LIB Therapeutics LLC (Industry)
Collaborators: Medpace, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LIB003-007
Record Dates: First submitted 2021-03-09; First posted 2021-03-15 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Cardiovascular Disease With Mention of Arteriosclerosis; Elevated Cholesterol; Familial Hypercholesterolemia
Keywords: lerodalcibep; PCSK9 inhibitor
MeSH Terms: conditions — Hypercholesterolemia; Hyperlipoproteinemia Type II

STUDY DESIGN:
Intervention Model Description: open label extension trial
Masking Description: lipids blinded to participant, investigator and sponsor at Day 1 only
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- LIB003 (lerodalcibep) (Experimental): 300 mg monthly (Q4W) by subcutaneous injection
  Interventions: Drug: lerodalcibep

INTERVENTIONS:
Drug: lerodalcibep — PCSK9 inhibitor
  Other Names: LIB003

SUMMARY:
The study is to assess the long-term safety, tolerability, and efficacy after 48 and 72 weeks with monthly (Q4W [<31 days]) dosing of subcutaneous (SC) LIB003 300 mg administered in patients with CVD or at high risk for CVD (including HoFH and HeFH) on stable diet and oral LDL-C lowering drug therapy who completed one of the LIB003 Phase 3 base studies.

DETAILED DESCRIPTION:
The population for this open-label study includes patients who successfully complete one of the randomized, controlled (placebo or comparator) blinded Phase 3 base studies (LIB003-003, LIB003-004, LIB003-005, LIB003-006, LIB003-008, LIB003-011 and LIB003-012). Patients will continue to maintain their existing oral lipid-lowering therapy (LLT).

Following completion of a base study and providing informed consent, patients will receive doses of LIB003 300 mg Q4W (<31 days) on Day 1 and Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, and 68. Patients will be seen in the clinic Q4W (<31 days) for at least the initial 12 weeks and then every 12 weeks (Weeks 24, 36, 48, 60, and 72) with the interim Q4W (<31 days) doses administered at home.

Patients may begin the OLE on the final visit of their prior study after completion of all requirements for that trial. Their lipids will remain blinded (to patient, study staff and sponsor) until week 4 to avoid any unblinding of the prior trial. Thereafter lipid results will be unblinded throughout the remainder of the 72 week trial.

ELIGIBILITY:
Inclusion Criteria:

* Successful completion 1 of one of the Phase 3 base studies LIB003-003, LIB003-004, LIB003-005, LIB003-006, LIB003-008, LIB003-011 and LIB003-012 without SAEs related to LIB003; or
* Provision of written and signed informed consent prior to any study-specific procedure;
* Female patients of childbearing potential must be using a highly effective form of birth control if sexually active and have a negative urine pregnancy test on Day 1 prior to dosing;
* Patient is willing to maintain appropriate diet and stable dose of current lipid-lowering therapy including statins, ezetimibe, bile acid sequestrants, niacin, bempedoic acid, bezafibrate or fenofibrate, and/or OM-3 compounds; and
* Patient is considered by the Investigator to be otherwise healthy,

Exclusion Criteria:

* Failure to complete a base Phase 3 (LIB003-003, LIB003-004, LIB003-005, LIB003-006, LIB003-008, LIB003-011 and LIB003-012) study and/or had an SAE that was related to study drug during the base Phase 3 study;
* Development since the final visit in the base Phase 3 (LIB003-003, LIB003-004, LIB003-005, LIB003-006, LIB003-008, LIB003-011 or LIB003-012) study of any concomitant clinical condition or acute and/or unstable systemic disease compromising patient inclusion, at the discretion of the Investigator,
* Use of prohibited oral lipid-lowering agents PCSK9 mAbs, mipomersen, lomitapide gemfibrozil (or bempedoic acid for LIB003, -011) following the base study or the use of PCSK9 short interfering ribonucleic acid (siRNA), or locked nucleic acid-reducing agents (LNA) within the last 6 months;
* Not available for protocol-required study visits or procedures, to the best of the patient's and Investigator's knowledge;
* Has any other finding which, in the opinion of the Investigator, would compromise the patient's safety or participation in the study;

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2020-12-03 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events as assessed by Medical Dictionary for Regulatory Activities as severe, moderate or mild after 48 and 72 weeks | 72 weeks
  Evaluation of Adverse Events based on MedRA based on ITT population

SECONDARY OUTCOMES:
Immunogenicity | 72 weeks
  Incidence of anti-drug antibodies
LDL Cholesterol reduction | 72 weeks
  Percent decrease in LDL-C from baseline of original study

CONTACTS AND LOCATIONS:
Overall Officials: David Kallend, MB BCh, Study Director — LIB Therapeutics
Locations (12):
- United States (4):
  - NorthShore University Health System, Evanston, Illinois
  - Sterling Research Group, Cincinnati, Ohio
  - The Lindner Research Center, Cincinnati, Ohio
  - Metabolic & Atherosclerosis Research Center (MARC), Cincinnati, Ohio
- G.B. Pant Institute of Postgraduate Medical Education & Research, New Delhi, India
- Israel (2):
  - Department of Medicine, Hadassah University Hospital, Jerusalem
  - Rabin Medical Center, Beilinson Hospital,, Petah Tikva
- Lipid Clinic, Oslo University Hospital, Oslo, Norway
- South Africa (2):
  - Carbohydrate and Lipid Metabolism Research Unit, Johannesburg, Gauteng
  - Division of Lipidology, Department of Medicine University of Cape Town, Cape Town, Western Province
- Turkey (Türkiye) (2):
  - Ege University Medical School, Izmir, Bornova
  - Afyonkarahisar Health Sciences University, Afyonkarahisar

IPD SHARING:
Plan to Share IPD: No